CLINICAL TRIAL: NCT02166034
Title: Healthy Gardens, Healthy Youth (HGHY): A People's Garden School Pilot Program
Brief Title: Effects of School Gardens on Children's Diet, Nutritional Knowledge, Etc.
Acronym: HGHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Washington State University (Other); University of Arkansas (Other); Iowa State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CN-CGP-11-0047
Record Dates: First submitted 2014-05-15; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-05

CONDITIONS: Dietary Habits
Keywords: children; fruit; vegetable; diet; school; garden
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- garden intervention (Experimental): Schools assigned to the garden intervention receive raised bed garden kits and access to a toolkit of garden-based curriculum
  Interventions: Behavioral: garden intervention
- Control (No Intervention): Wait-list control (no garden intervention + lessons) until end of the study.

INTERVENTIONS:
Behavioral: garden intervention — The intervention includes raised bed garden kits for participating classes as well as access to garden-based curriculum.
  Arms: garden intervention

SUMMARY:
The purpose of this study is to determine whether school gardens influence children's dietary intake, nutritional knowledge, and other outcomes.

DETAILED DESCRIPTION:
Schools in New York, Washington State, Iowa, and Arkansas were randomly assigned to receive school gardens and associated curriculum or to serve on the wait list control group that received gardens and curriculum at the end of the 2-year study. Baseline data were collected in Fall 2011. Garden interventions began in Spring 2012. Follow-up data were collected at 6, 12, 18 months following baseline data collection.

ELIGIBILITY:
Inclusion Criteria:

* Schools had at least 50% of enrolled children qualifying for free + reduced price meals (FRPM)
* Schools did not already have a school garden.

Exclusion Criteria:

none.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3531 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
change in fruit + vegetable intake at school | change from baseline to follow-up at 6, 12, 18 months
  Children's lunch trays are photographed before and after lunch for 3 days at each wave of data collection. Digital Food Image Analysis software computes grams of fruit and grams of vegetables consumed for each pair of lunch tray photos.

SECONDARY OUTCOMES:
Garden Intervention Fidelity | At 3 garden intervention time points -- 6, 12, 18 months after baseline
  fruit + vegetables planted, harvested; methods of fruit and vegetable distribution; and garden-based lessons delivered to the class are measures at each wave of data collection from Fall 2011 to Spring 2013.
change fruit & vegetable consumption at home | change from baseline (Fall 2011) to follow-up at 6 months, 12 months, 18 months.
change in Nutritional Knowledge | change from baseline to follow-up at 6, 12, 18 months
  In the classroom, children complete a 7-item multiple choice questionnaire developed by the Healthy Gardens, Healthy Youth curriculum development team. The questionnaire includes items about plant science (e.g., Which part of the plant uses the sun's energy to make food? root, stem, leaf, flower) and nutrition (e.g., Which nutrient supplies our bodies with energy? fiber, carbohydrates, water, vitamins). Data represent the number of correct answers.
change in Science Technology Engineering Math (STEM) self efficacy | change from baseline (Fall 2011) to follow-up at 6, 12, 18 months.
  In the classroom, children complete a 15-item questionnaire, derived from the Science Process Skills Inventory (SPSI) (Arnold & Bourdeau, 2009) and the Iowa 4-H Science Youth Self-Assessment (Staker, 2011). Items include, for example: "I can do an experiment to answer a question" and "I can develop a plan for a good garden I want to plant" with response options "Disagree." "Not Sure." or "Agree" denoted 1, 2, or 3 respectively. The STEM self-efficacy score range is thus 15-45, with higher scores indicating that participant has stronger positive beliefs in their abilities to use STEM to solve problems.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Wells, PhD, Study Director — Cornell University
Locations (4):
- United States (4):
  - Schools in Arkansas, Little Rock, Arkansas
  - Schools in Iowa, Osceola, Iowa
  - Schools in New York State, Ithaca, New York
  - Schools in Washington State, Tacoma, Washington

REFERENCES:
- [Derived] Wells NM, Meyers BM, Todd LE, Henderson CR Jr, Barale K, Gaolach B, Ferenz G, Aitken M, Tse CC, Pattison KO, Hendrix L, Carson JB, Taylor C, Franz NK. The carry-over effects of school gardens on fruit and vegetable availability at home: A randomized controlled trial with low-income elementary schools. Prev Med. 2018 Jul;112:152-159. doi: 10.1016/j.ypmed.2018.03.022. Epub 2018 Apr 5. PMID 29627512